CLINICAL TRIAL: NCT03266835
Title: A Multinational, Single-Arm Pivotal Study to Assess the Performance Rate Of SoundBite™ Active Wire for PEripheral Chronic Total Occlusion Recanalization (PROSPECTOR)
Brief Title: SoundBite™ Crossing System Pivotal Peripheral CTO Crossing Study
Acronym: PROSPECTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SoundBite Medical Solutions, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry); Prairie Vascular Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAP-PER-2017-01
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Chronic Total Occlusion of Arteries of the Extremities
Keywords: Chronic Total Occlusion; Peripheral; SoundBite™ Crossing System; CTO; intra-luminal; Active wire; Device; Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SoundBite™ Crossing System - Peripheral (Other): This is a multinational, single-arm, pivotal trial assessing the efficacy and safety of the SoundBite™ Crossing System with subjects diagnosed with de novo infrainguinal arterial chronic total occlusion(s).
  Interventions: Device: SoundBite™ Crossing System - Peripheral

INTERVENTIONS:
Device: SoundBite™ Crossing System - Peripheral — SoundBite™ Crossing System consisting of the SoundBite™ Console and SoundBite™ Active Wire 18. The Investigator may use the SoundBite™ Active Wire during the procedure to cross the proximal aspect and/or to cross multiple lesions.

SUMMARY:
This study is aimed at demonstrating the efficacy and safety of the SoundBite™ Crossing System-Peripheral. The study is intended to demonstrate that the SoundBite™ Crossing System can facilitate the passage of either devices intended to treat a chronic total occlusion (CTO) or additional crossing devices through an infrainguinal CTO into the true lumen.

DETAILED DESCRIPTION:
This is a multinational, single-arm, pivotal trial assessing the efficacy and safety of the SoundBite™ Crossing System - Peripheral. The enrollment will consist of up to 100 patients meeting the inclusion/exclusion criteria in order to obtain 90 evaluable patients for efficacy and safety analysis. The primary endpoints will be compared to literature-based performance goals to establish study success.

Objective Performance Goals (OPG) have been obtained from a literature based review. Reports published in the past 10 years were reviewed for both safety and effectiveness in crossing infrainguinal CTO. The studies reviewed generally have one primary composite safety endpoint and one primary efficacy endpoint. Some studies have performed formal hypothesis testing versus a pre-specified performance goal for one or both endpoints.

ELIGIBILITY:
General Inclusion Criteria:

1. Has symptomatic chronic limb ischemia, requiring treatment of an in:frainguinal artery
2. Has Rutherford Clinical Category of 2-5
3. Is ≥ 18 years old
4. Has life expectancy > 1 year
5. Is able and willing to provide written informed consent prior to study procedure

Angiographic Inclusion Criteria:

Unless otherwise specified, the Investigator performing the procedure bases angiographic inclusion on visual determination of qualification imaging taken at time of procedure.

Subject must meet ALL the following angiographic inclusion criteria:

1. Has evidence of a clinically significant de novo CTO located in a peripheral vessel below the infrainguinal ligament confirmed by angiography at time of procedure.
2. Notwithstanding criteria 1, multilevel CTOs are included as long as the total length from the beginning of the most proximal total occlusion to the end of the most distal total occlusion is less than 40 cm.
3. 100% stenosis by visual estimate of angiography at time of procedure.
4. Has target limb with at least one patent (<50% stenosis) run-off vessel confirmed by angiography or magnetic resonance angiography at time of procedure.

General Exclusion Criteria:

1. Has had a previous peripheral bypass that includes the target vessel.
2. Has had a previous intervention on the target CTO (e.g., angioplasty, stent placement), including previous attempt at time of index procedure.
3. History of any vascular procedure on the index limb within the last 30 days requiring clinically driven re-intervention.
4. Has an active infection in the target limb.
5. Subject has any planned major surgical or interventional procedure within 30 days after the study procedure.
6. Has received a kidney transplant.
7. Glomerular Filtration Rate (GFR) of less than 40.
8. Unstable coronary artery disease or other uncontrolled comorbidity.
9. Myocardial infarction or stroke within 2 months prior to baseline evaluation.
10. Subject has positive pregnancy test result in women of child bearing potential or is breast-feeding.
11. Participation in any study of an investigational device, medication, biologic, or other agent during study or within 30 days prior to enrollment that is either a cardiovascular study or could, in the judgment of the investigator, affect the results of this study.
12. Subject in whom antiplatelet, anticoagulant therapy is contraindicated
13. Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 100,000/ml or known coagulopathy.
14. Known, untreated allergy to contrast agents or medications used during or subsequent to endovascular intervention. Patients with aspirin allergy that have been desensitized are not excluded.
15. History of heparin-induced thrombocytopenia (HIT) that cannot be treated with direct thrombin inhibitors.
16. Any thrombolytic therapy within two weeks prior to enrollment.
17. Psychiatric disorder which in the judgment of the investigator could interfere with provision of informed consent, completion of tests, therapy, follow-up or general study compliance

    Angiographic Exclusion Criteria

    Unless otherwise specified, the Investigator performing the procedure bases angiographic exclusion on visual determination of qualification imaging taken up to 6 months prior to procedure and/or imaging taken at time of procedure. Subject is excluded if ANY of the following angiographic exclusion criteria is met:
18. Has significant stenos is or occlusion of inflow tract ( upstream disease) unsuccessfully treated at time of index procedure or presenting symptoms such as embolism confirmed by angiography.
19. Has in a native vessel, a previously stented segment separated by < 3 cm of angiographically normal vessel from the target CTO.
20. CTOs lacking at least one patent target distal artery (::;SO% diameter stenosis).
21. Has an acute or sub-acute intraluminal thrombus within the target vessel.
22. Aneurysm distal to puncture access site at least twice the reference vessel diameter, located in the index vessel, abdominal aorta, iliac or popliteal.
23. Has perforation, dissection or other injury of the access site or index vessel requiring stenting or surgical intervention prior attempting crossing of the target lesion with SoundBite™ Crossing System.
24. Clinical/angiographic evidence of distal embolization in the index extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Technical Device Success | Day 1
  Ability to facilitate treatment of the target lesion by allowing additional crossing and/or treatment devices to cross the CTO
Freedom from SoundBite™ Crossing System related MAEs at 30 days post procedure | up to Day 30
  MAEs defined as:
  * Cardiovascular related deaths
  * Unplanned, index limb amputation
  * Dissection of grade C or greater that require an intervention to resolve
  * Symptomatic distal embolization, defined as clinical signs or symptoms of distal emboli detected in the treated limb distal to the treated lesion after the index procedure or noted angiographically after the index procedure, and requiring mechanical or pharmacologic means to improve flow

SECONDARY OUTCOMES:
Procedural success | Day 1
  Achievement of Technical Success together with post-procedural patency. Post-procedural patency is defined as less then or equal to 50% residual percent diameter stenosis assessed by visual estimate at the end of revascularization procedure
Clinical Success | Up to Day 30
  Achievement of Procedural Success as well as freedom from SoundBite™ Crossing System related MAEs at 30 days
Penetration ≥ 0.5 cm | Day 1
  Ability of the SoundBite™ Crossing System to penetrate ≥ 0.5 cm of any segment of the CTO
Fully traverse | Day 1
  Ability of the SoundBite™ Crossing System to fully traverse the CTO with entry into the distal true lumen without the need for additional guidewires and/or re-entry devices
Freedom from any SoundBite™ Crossing System related Adverse Events | Up to Day 30
  Freedom from any SoundBite™ Crossing System related Adverse Events

CONTACTS AND LOCATIONS:
Locations (2):
- UNC Rex Healthcare, Raleigh, North Carolina, United States
- CHUM-Hôtel-Dieu du Centre Hospitalier Universitaire de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No